CLINICAL TRIAL: NCT01655524
Title: The Impact of Routine Administration of Aminophylline Following Regadenoson According to the ASSUAGE Protocol on the Accuracy of Regadenoson Stress Myocardial Perfusion Imaging: A Single-Blinded Cross-Over Clinical Trial
Brief Title: The Impact of the Routine Aminophylline Administration Following Regadenoson Stress on SPECT Myocardial Perfusion
Acronym: ASSUAGE-MPI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to nationwide shortage of Aminophylline. No subjects enrolled.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ASSUAGE-MPI Trial
Record Dates: First submitted 2012-07-26; First posted 2012-08-02 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
Keywords: Regadenoson; Aminophylline; ASSUAGE; Myocardial Perfusion Imaging (MPI)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aminophylline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ASSUAGE Protocol (Experimental): There is only one arm in this cross-over design trial. Patients who had a standard regadenoson stress test will be invited to enroll in the study. All enrolled subjects will undergo an investigational (ASSUAGE) regadenoson stress test. Imaging scans from the same patients (scan 1 and scan 2) will be compared.
  Interventions: Drug: ASSUAGE Protocol

INTERVENTIONS:
Drug: ASSUAGE Protocol — 75 mg of aminophylline injected intravenously 90 seconds following the radioisotope injection in the setting of regadenoson nuclear stress test of the heart.
  Other Names: Aminophylline

SUMMARY:
The investigators developed a modified regadenoson nuclear stress test of the heart that incorporates an aminophylline injection following regadenoson (The ASSUAGE protocol). The modified (ASSUAGE) protocol has been associated with fewer side effects and was better tolerated by patients.

This study will investigate whether the modified regadenoson stress protocol (ASSUAGE) produces blood flow pattern to the heart similar to that of a standard regadenoson stress protocol. In proven to be the case, the ASSUAGE protocol has the potential to be used on a wide scale instead of the current standard protocol.

DETAILED DESCRIPTION:
Patients who had regadenoson stress nuclear stress test of the heart will be invited to return to undergo a modified nuclear stress using the modified (ASSUAGE) protocol. Images from the original scan will be compared to those from the second scan to determine whether the blood flow pattern is similar between the two scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a qualifying regadenoson stress myocardial perfusion imaging (regadenoson nuclear stress test).

Exclusion Criteria:

* inability to provide an informed consent
* known allergic reaction to aminophylline or regadenoson
* systolic blood pressure < 90 mmHg
* unstable abnormal heart rhythm
* pulmonary edema
* acute coronary symptoms, myocardial infarction within 48 hours
* active dipyridamole, aminophylline or theophylline use
* pregnancy
* any contraindication to aminophylline according to the drug's package insert: uncontrolled seizure disorder, sepsis with multi-organ failure and liver impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Summed Difference Score (SDS); a measure of size and severity of ischemia (heart muscle in jeopardy) detected with regadenoson nuclear stress of the heart (standard vs. ASSUAGE protocol). | The second (investigational) stress will be performed within 4 weeks from the intial one.
  The SDS produced with standard protocol will be compared to SDS produced with the modified (ASSUAGE) protocol. The study is set out to demonstrate that there is no significant difference in SDS between the two protocols within the same patients.

SECONDARY OUTCOMES:
Agreement rate in the SDS burden category (normal/mild, moderate or severe) | within 4 weeks
  Agreement rate in the SDS burden category (normal/mild, moderate or severe)between scan 1 and scan 2 will be compared to the agreement rate between 2 sets of images from scan 1. The study is set out to demonstrate that these agreement rates are not significantly different.

OTHER OUTCOMES:
Agreement rate in the size of blood flow abnormality category (none/small, moderate or large) | within 4 weeks
  Agreement rate in the SDS burden category (normal/mild, moderate or severe)between scan 1 and scan 2 will be compared to the agreement rate between 2 sets of images from scan 1. The study is set out to demonstrate that these agreement rates are not significantly different.

CONTACTS AND LOCATIONS:
Overall Officials: Rami Doukky, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States